CLINICAL TRIAL: NCT06799286
Title: An Open-label, Single-arm, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BMS-986489 (BMS-986012 + Nivolumab Fixed Dose Combination) in Chinese Participants With Relapsed/Refractory Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BMS-986489 in Chinese Participants With Relapsed/Refractory Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA245-0002
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: BMS-986489; atigotatug; BMS-986012; SCLC; fucosyl-GM1
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BMS-986489 (Experimental)
  Interventions: Drug: BMS-986489

INTERVENTIONS:
Drug: BMS-986489 — Specified dose on specified days

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, and preliminary efficacy of BMS-986489 in Chinese participants with R/R SCLC (Relapsed/Refractory Small Cell Lung Cancer).

ELIGIBILITY:
Inclusion Criteria:

- Participants must have histologically or cytologically documented SCLC (small cell lung cancer). Participants with either limited or extensive disease stage at the initial diagnosis, who have received at least one prior line of systemic therapy, are eligible.

i) For initial limited stage (LS) SCLC:.

A. Those who progressed or recurred after more than 6 months treatment-free interval following treatment of curative surgical resection, systemic therapy, or radiotherapy, and subsequently received at least one line of systemic therapy to treat the recurrence or progression, and then progressed, or were intolerant to the prior systemic therapy per the assessment of investigators, these participants will be eligible, or

B. Who progressed or recurred within 6 months after treatment of curative surgical resection, systemic therapy, or radiotherapy, no matter if these participants have received subsequent systemic therapy, these participants will be eligible.

ii) For initial extensive stage (ES) SCLC, participants must have received at least one line of platinum-based systemic therapy (with/without immunotherapy), and then progressed, or been intolerant to the prior systemic therapy per the assessment of investigators.

A. Note: 1) For ES-SCLC with only one line of platinum-based regimen as well as chemotherapy-free interval is more than 6months when progression, only when participants refuse or are ineligible for re-treatment with platinum-based doublet per the assessment of investigators, these participants will be eligible. 2) If participants receive re-treatment with a platinum-based regimen, it is considered a second line of therapy.

* Participants must have a life expectancy of ≥12 weeks.
* Participants must have at least 1 measurable lesion outside the central nervous system (CNS) by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.

Exclusion Criteria:

* Untreated symptomatic CNS metastases.
* Leptomeningeal disease.
* Pleural effusion which cannot be controlled with appropriate interventions.
* Malignancy-related superior vena cava syndrome.
* Participants with an active, known or suspected, autoimmune disease.
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to first study treatment.
* Unresolved toxicity from prior anti-tumor therapy.
* Prior treatment with an anti-fuc-GM1 therapy or any other drug specifically targeting fuc-GM1.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-05-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 12 months after last participant's first treatment
Number of participants with Serious AEs (SAEs) | Up to 12 months after last participant's first treatment
Number of participants with AEs leading to discontinuation of study treatment | Up to 12 months after last participant's first treatment
Number of participants with select AEs | Up to 12 months after last participant's first treatment
Number of participants with immune-mediated AEs (IMAEs) | Up to 12 months after last participant's first treatment
Number of deaths | Up to 12 months after last participant's first treatment
Number of participants with laboratory abnormalities | Up to 12 months after last participant's first treatment
Maximum observed concentration (Cmax) for BMS-986012 | Up to 12 months after last participant's first treatment
Time of maximum observed concentration (Tmax) for BMS-986012 | Up to 12 months after last participant's first treatment
Trough observed plasma concentration (Ctrough) for BMS-986012 | Up to 12 months after last participant's first treatment
Concentration at the end of a dosing interval (Ctau) for BMS-986012 | Up to 12 months after last participant's first treatment
Average concentration over a dosing interval ([AUC(TAU)/TAU]) (Cavg(TAU)) for BMS-986012 | Up to 12 months after last participant's first treatment
Area under the concentration-time curve within one dosing interval (AUC(TAU)) for BMS-986012 | Up to 12 months after last participant's first treatment
Total body clearance (CLT) for BMS-986012 | Up to 12 months after last participant's first treatment
Observed concentration at end of infusion (Ceoi) for BMS-986012 | Up to 12 months after last participant's first treatment

SECONDARY OUTCOMES:
Number of participants with anti-drug antibodies (ADAs) to BMS-986012 | Up to 12 months after last participant's first treatment
Number of participants with ADAs to nivolumab | Up to 12 months after last participant's first treatment
Ctrough for nivolumab | Up to 12 months after last participant's first treatment
Ceoi for nivolumab | Up to 12 months after last participant's first treatment
Overall Response (OR) | Up to 12 months after last participant's first treatment
  Achievement of best response of complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, assessed by the investigator.
Disease Control (DC) | Up to 12 months after last participant's first treatment
  Achievement of best response of CR or PR or stable disease (SD) using RECIST v1.1 criteria, assessed by the investigator.
Duration of Response (DOR) | Up to 12 months after last participant's first treatment
  Time from first response (CR or PR) to first documented disease progression by investigator or death, whichever occurs first. For participants who did not have an event, the DOR will be censored on the date of their last tumor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- China (5):
  - Local Institution - 0004, Beijing, Beijing Municipality
  - Local Institution - 0003, Jinan, Shandong
  - Local Institution - 0001, Linyi, Shandong
  - Local Institution - 0005, Hangzhou, Zhejiang
  - Local Institution - 0002, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html